CLINICAL TRIAL: NCT06602076
Title: Developing an Empowerment Theory-Based Smoking Cessation Intervention for People With High Levels of Social Stress
Brief Title: Developing Empowering Smoking Cessation
Acronym: ECHO
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17583; 1R34DA060534-01A1 (NIH)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Smoking Cessation
Keywords: tobacco use; smoking cessation; stress; social support; community engaged
MeSH Terms: conditions — Smoking Cessation; Tobacco Use

STUDY DESIGN:
Intervention Model Description: In a 2-arm, 12-week pilot randomized controlled trial (RCT) with Week 24 follow up, N=50 adults willing to quit smoking from Oklahoma (OK) and the San Joaquin Valley (SJV) in California will be randomized to receive either the NCI's quitSTART smoking cessation smartphone app and free nicotine replacement therapy (NRT; control, n=25), or quitSTART and NRT plus ECHO, which includes online community-serving volunteer activities (≥4 sessions) and a digital hub (Reddit) to foster social support across sites.
Who Masked: Outcomes Assessor
Masking Description: Blinding participants will not be possible because participants will be able to tell if they are in the treatment group versus control group due to the volunteer activities in the treatment group and absence of such activities in the control group. Investigators will remain blinded to the group assignments. Randomization will use a centralized and automated system to ensure allocation concealment from outcomes analysts. If manual allocation is required, sequentially numbered, opaque, sealed envelopes will be utilized to maintain allocation concealment and managed internally at OU. Additionally, the following blinded outcome assessment procedures are planned: Outcome assessors will be a separate and unique team from those managing allocation and tracking of participants during the research activities; Participants will be assigned unique codes that do not reveal their identity and group to the outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Receive standard smoking cessation treatment in the form of the NCI's quitSTART smoking cessation smartphone app and free over-the-counter nicotine replacement therapy provided by mail, plus participate in online community-serving volunteer activities (≥4 sessions) and a digital hub (Reddit) to foster social support across sites.
  Interventions: Behavioral: ECHO (Empowering Our Community & Health Outcomes)
- Control (No Intervention): Receive standard smoking cessation treatment in the form of the NCI's quitSTART smoking cessation smartphone app and free over-the-counter nicotine replacement therapy provided by mail.

INTERVENTIONS:
Behavioral: ECHO (Empowering Our Community & Health Outcomes) — Additive intervention design wherein study participants receive remotely-delivered standard smoking cessation support (i.e., behavioral support plus nicotine replacement therapy) and engage in community-serving volunteer activities.
  Arms: Treatment

SUMMARY:
Problem: Despite encouraging use declines in the U.S. population, tobacco is still a leading cause of preventable disease and death. Current cessation treatments have limited success; two-thirds relapse within 6 months of a quit attempt. Existing smoking cessation interventions overwhelmingly focus on within-person processes of behavior change rather than socioenvironmental influences on cessation success. Cessation interventions based on evidence linking social stress to increased nicotine dependence and relapse risk are needed to address the stressors people who smoke encounter while navigating their social environments (i.e., social stress). Effective empowering approaches for infectious disease prevention and youth tobacco use suggest that Empowerment Theory may also enhance smoking cessation assistance for people experiencing high levels of social stress.

Hypothesis: Our hypothesis is that when people participate in community-serving volunteer activities, they may also experience cognitive and behavioral changes (i.e., enhanced stress coping, social support, self-worth, prosociality) that ameliorate the effects of social stress, thereby supporting smoking cessation.

Importance: Empowerment Theory-informed health behavior change approaches have worked for infectious disease prevention and youth tobacco interventions. Our pretest (N=20; Oklahoma) demonstrated the feasibility and acceptability of volunteer activity participation as an adjunct to standard smoking cessation treatment. This novel smoking cessation intervention uses an innovative, theory-based, local-yet-scalable approach to enhance individual outcomes through community engagement. To ensure scalability and accessibility of this remotely delivered intervention, we will utilize the NIH-supported Dissemination and Implementation (D&I) science framework, the Practical, Robust Implementation and Sustainability Model (PRISM), which is the contextually expanded version of RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance). This project will advance efforts to understand and address high tobacco use among people experiencing high levels of social stress and will inform a future R01 application for a fully-powered, multi-site RCT of ECHO aiming to end tobacco use across the U.S. while supporting community connectedness.

DETAILED DESCRIPTION:
Specific Aims

Aim 1 (Inform): Prioritize factors associated with smoking cessation for people with high levels of social stress to inform volunteer activity protocol development for ECHO. We will use smartphone-administered ecological momentary assessment (EMA) to observe a 28-day naturalistic cessation attempt with N=60 adults with high levels of social stress recruited nationally. We will assess daily cessation-related experiences and behaviors, including evidence-based cessation factors (e.g., stress coping). These factors likely fluctuate within and across days, requiring EMA. Hypothesis: Stress coping, social support, self-worth, and prosociality will be associated with within- and day-level smoking abstinence, with largest effect sizes for social support and self-worth.

Aim 2 (Develop): Develop volunteer activity protocols likely to maximize smoking cessation success for people with high levels of social stress. With findings on prioritized cessation factors from Aim 1, our community partners, and our pretesting experience, we will develop a set of online volunteer activities that support participants' communities and harness key evidence-based cessation-promoting factors. Activities will be iteratively tested and refined with feedback from N=12 adults with high levels of social stress and volunteer activity facilitators in OK and SJV. These will form the basis of ECHO's refined core protocol that can be readily adapted in future intervention iterations.

Aim 3 (Pilot): Determine the feasibility, acceptability, and associations with quit self-efficacy and motivation of the developed ECHO protocol in two pilot sites. In a 2-arm, 12-week pilot randomized controlled trial (RCT) with Week 24 follow up, N=50 adults from OK and SJV with high levels of social stress who are willing to quit smoking will be randomized to receive either the NCI's quitSTART smoking cessation smartphone app46 and free nicotine replacement therapy (NRT; control, n=25), or quitSTART and NRT plus ECHO, which includes online community-serving volunteer activities (≥4 sessions) and a digital hub (Reddit) to foster social support across sites. Key feasibility outcomes assessed at Week 12 include: intervention acceptability, quitSTART app engagement, NRT adherence, quit self-efficacy and motivation, smoking behavior, and cessation-promoting factors that we aim to activate with the volunteer activity protocols. Community partner outcomes will include volunteer hours and organizational visibility as assessed by participant records and key informant interviews. We will identify characteristics across volunteer activity protocols that best activated cessation-related factors.

ELIGIBILITY:
Inclusion/exclusion criteria (All Aims):

* Sexual and/or gender minority (SGM)-identified
* Adults (i.e., ≥ 18 years old)
* Currently smoking cigarettes
* Living in a high stigma environment in the U.S.
* Able to read English at > 6th-grade level

Individuals with serious psychological distress (i.e., score of 13 ≥ 18 on the Kessler PD Scale-6 19) will be excluded from all Aims because of likelihood of functional impairments that substantially interfere with one or more major life activities.

Aim 3 (Pilot RCT) inclusion criteria will be:

* (1) ≥ 18 years old
* (2) sexual and/or gender minority-identified (see definition above)
* (3) living in Oklahoma or one of the 8 counties in San Joaquin Valley, California (verified by address)
* (4) a current cigarette smoker (see definition above)
* (5) willing to quit smoking within 30 days of enrollment (see definition above)
* (6) own a smartphone
* (7) ability to read English at > 6th-grade level (see definition above)
* have no NRT contraindications
* (8) ≥ weekly internet access
* (9) willing and able to participate in SGM-serving volunteer activities.

Aim 3 (Pilot RCT) exclusion criteria: Individuals will be excluded if currently using other smoking cessation treatments.

Sexual minority identity will be indicated by selecting any non-heterosexual response option(s) from: Heterosexual (Straight); Gay or Lesbian; Bisexual; Something else (please state)." Participants will indicate the sex assigned on their birth certificate (i.e., natal sex). Gender minority identity will be indicated by "Trans male/Trans man;" "Trans female/Trans woman;" "Gender queer/Gender non-conforming;" "Different identity (please state)" or a binary identity (male or female) non-concordant with natal sex. Current cigarette smoking will be indicated by ≥100 lifetime cigarettes and currently smoking cigarettes "every day" or "some days". High SGM stigma states are defined as the 22 states wherein ˂60% of the population 'thinks that homosexuality should be accepted'.21 High SGM stigma municipalities are defined as one of the 246 U.S. municipalities (out of the 496 scored from all U.S. states) that scored below the median (71) on the HRC Municipal Equality Index. Willingness to quit smoking will be assessed with a single item: "Are you willing to quit smoking cigarettes within 30 days after enrolling in this study? (yes/no)". To be classified as 'ready to quit smoking,' participants will report readiness to quit in the next 30 days and at least 1 past-year quit attempt (i.e., in the "Preparation" stage of change).

An equal number of female and male participants (i.e., natal sex) will be recruited so as to examine sex as a biological factor. Recruitment targets will aim to reflect the racial/ethnic composition of the populations from which the samples are drawn.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Retention | 12 weeks
  BENCHMARK:
  Retention at week 12 (minimum 80%)
Intervention feasibility | 12 weeks
  The following post-intervention outcome will be assessed at Week 12: Overall intervention feasibility will be assessed by the Weiner scale (2017), which has four 5-point Likert-scale questions; higher score indicates greater feasibility.
  BENCHMARK:
  Intervention feasibility at Week 12 (70% or more of participants with an average score of 4 or greater on each scale).
Intervention acceptability | 12 weeks
  The following post-intervention outcome will be assessed at Week 12: Overall intervention acceptability will be assessed by the Weiner scale (2017), which has four 5-point Likert-scale questions; higher score indicates greater acceptability.
  BENCHMARK:
  Intervention acceptability at Week 12 (70% or more of participants with an average score of 4 or greater on each scale).
Intervention appropriateness | 12 weeks
  The following post-intervention outcome will be assessed at Week 12: Overall intervention appropriateness will be assessed by the Weiner scale (2017), which has four 5-point Likert-scale questions; higher score indicates greater appropriateness.
  BENCHMARK:
  Intervention appropriateness at Week 12 (70% or more of participants with an average score of 4 or greater on each scale).

SECONDARY OUTCOMES:
Self-reported smoking abstinence assessed at Week 12 | 12 weeks
  -Self-reported 7-day Point Prevalence Abstinence (PPA)
Self-efficacy asssessed at Week 12 | 12 weeks
  -Self-Efficacy Scale/Confidence (SESC)
Motivation to quit smoking assessed at Week 12 | 12 weeks
  -Motivation to change (Stages of Change [SoC] scale)
Smoking intensity assessed at Week 12 | 12 weeks
  -Smoking intensity will be assessed by past-week smoking days and past-week cigarettes per smoking day.
Cessation Treatment Engagement assessed at Week 12 | 12 weeks
  -Engagement with smoking cessation treatment will be the number of days the participant opened the quitSTART app during the 12-week intervention period according to objective -tracking of app feature use. Greater number of days indicates greater engagement.

OTHER OUTCOMES:
Self-reported smoking abstinence assessed at Week 24 | 24 weeks
  -Self-reported 7-day Point Prevalence Abstinence (PPA)
Smoking intensity assessed at Week 24 | 24 weeks
  -Smoking intensity will be assessed by past-week smoking days and past-week cigarettes per smoking day.
Motivation to quit smoking assessed at Week 24 | 24 weeks
  -Motivation to change (Stages of Change [SoC] scale)
Self-efficacy asssessed at Week 24 | 24 weeks
  -Self-Efficacy Scale/Confidence (SESC)

CONTACTS AND LOCATIONS:
Overall Officials: Julia M McQuoid, PhD, Principal Investigator — Associate Professor

IPD SHARING:
Plan to Share IPD: Yes
All dataset(s) that can be shared will be deposited in the Inter-university Consortium for Political and Social Science Research (ICPSR) data archive; a unit within the Institute for Social Research at the University of Michigan with offices in Ann Arbor. Should availability of this Consortium change during the course of the project an NIH-supported data repository will be used. The ICPSR data archive provides metadata, persistent identifiers (i.e., Digital Object Identifiers or DOI) and long-term access. ICPSR hosts data in a repository with powerful search capabilities. This repository is supported by the University of Michigan's Institute for Social Research and datasets are available through a request process.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available as soon as possible or (at the latest) at the time of associated publication. The duration of preservation and sharing of the data will be a minimum of five years after the end of the funding period but is anticipated to continue in perpetuity.
Access Criteria: Access to data will be controlled as restricted-use. Given the sensitive information (I.e., enables the potential identification of respondents from rural settings through inference) the dataset, de-identified individual participant-level data will be made available in the ICPSR repository, which restricts access to qualified investigators with an appropriate research question who sign a data use agreement and undergo an approval process.
URL: http://www.icpsr.umich.edu/web/pages/